CLINICAL TRIAL: NCT00926302
Title: A Randomized, Single, Two-Way Crossover Pivotal Study to Assess the Bioequivalence Study of Levetiracetam vs. Keppra Administered Under Fasting Conditions to Healthy Adult Subject
Brief Title: A Bioequivalence Study of Levetiracetam Versus Keppra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: I-Shin Shiah/The Head of Department of Psychiatry, Tri-Service General Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MCPE08034M1; TSGHIRB097-02-006; C159
Record Dates: First submitted 2009-06-18; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: The bioequivalence of Levetiracetam vs. Keppra; volunteer
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test drug (Experimental): Levetiracetam one period
  Interventions: Drug: Levetiracetam (Lotus Pharmaceutical Co.,Ltd.)
- Reference drug (Active Comparator): Keppra one period
  Interventions: Drug: Keppra (Levetiracetam - USB SA Pharma Sector)

INTERVENTIONS:
Drug: Levetiracetam (Lotus Pharmaceutical Co.,Ltd.) — Levetiracetam 500mg/tablet Oral once
  Other Names: The test drug Levetiracetam is no brand name.; Manufacturer:Lotus Pharmaceutical Co.,Ltd.
  Arms: Test drug
Drug: Keppra (Levetiracetam - USB SA Pharma Sector) — Levetiracetam 500mg/tablet oral once
  Other Names: Keppra; Manufracturer:USB SA Pharma Sector
  Arms: Reference drug

SUMMARY:
The purpose of this study is to assess the bioequivalence of Levetiracetam versus Keppra administered under fasting conditions to healthy adult subjects.

DETAILED DESCRIPTION:
This study is a randomized, single, two-way crossover pivotal study. The pharmacokinetic blood samples and vital signs were obtained before and after administration at scheduled intervals as indicated in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent before enrollment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
2. Healthy adult male, aged between 20 and 40 years old.
3. Body Mass Index between 18.5 and 25 (inclusive).
4. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest x-ray and electrocardiogram.
5. No significant deviation from normal biochemistry examination.
6. No significant deviation from normal hematology examination.
7. No significant deviation from normal urinalysis examination.

Exclusion Criteria:

1. History of drug or alcohol abuse within the past year.
2. Medical history of severe drug allergy or sensitivity to analogous drug.
3. Evidence of acute or chronic disease or having undergone surgery from 4 weeks prior to Period I dosing.
4. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology.
5. Ongoing peptic ulcer and constipation.
6. Planned vaccination during the time course of the study.
7. Taking any clinical investigation drug from 2 months prior to Period I dosing.
8. Use of any medication, including herb medicine or vitamins from 4 weeks before the study.
9. Blood donation of more than 500 mL within the past 3 months.
10. A positive Hepatitis B surface antigen or positive Hepatitis C antibody result.
11. A positive test for HIV antibody.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the bioequivalence | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: I-Shin Shiah, M.D., Principal Investigator — Tri-Service General Hospital